CLINICAL TRIAL: NCT01457066
Title: Culturally Sensitive Intervention to Improve Retention in HIV Care for Latino MSM
Acronym: PODER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, William Cunningham, Prinicipal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH089719-01A1 (NIH)
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): This group will receive the peer navigator intervention.
  Interventions: Behavioral: Peer Navigator Intervention
- Control (No Intervention): This group will receive usual care.

INTERVENTIONS:
Behavioral: Peer Navigator Intervention — Peer navigators will teach HIV retention and linkage skills and knowledge using group-based as well as one-on-one, peer-based learning approaches.
  Arms: Intervention

SUMMARY:
The goal of this proposal is to culturally adapt and tailor an existing, theory-based intervention, using state-of-the-art methods designed to maximize cultural sensitivity, feasibility and acceptability to HIV+ Latino MSM, and to test it in a small randomized controlled trial (n=60 intervention; n=60 control).

DETAILED DESCRIPTION:
While early receipt of and adherence to antiretroviral therapy are critical for effective HIV treatment, engagement with and retention in HIV care are essential first steps. Retention in HIV care is particularly important for traditionally disadvantaged groups, such as Latino MSMs, who are over-represented in the HIV epidemic. HIV+ Latino MSM therefore urgently need interventions to improve their retention in HIV care, which may be affected by a number of culture-specific factors. The goal of this proposal is to culturally adapt and tailor an existing, theory-based intervention, using state-of-the-art methods designed to maximize cultural sensitivity, feasibility and acceptability to HIV+ Latino MSM, and to test it in a small randomized controlled trial (n=60 intervention; n=60 control). The study will be conducted among insufficiently retained HIV+ Latino MSM at AltaMed, the largest provider of HIV medical services for Latinos in Los Angeles. The proposed intervention is designed to retain participants in HIV care by addressing barriers to and facilitators of HIV care salient to Latinos, using group-based as well as one-on-one, peer-based learning approaches.

ELIGIBILITY:
Inclusion Criteria include: 1) being HIV+; 2) > 18 years old; 3) male; 4) fluent in Spanish; 5) self-identify as having Latino or Hispanic ethnicity; 6) Self-identify as gay or as ever having sex with men; 7) Must have scheduled visit with AltaMed in the prior 12 months and have a) fewer than one visit in the prior four months or b) detectable viral load

Exclusion Criteria include 1) not having a scheduled visit with AltaMed in the prior 12 months and having a) more than one visit in the prior four months or b) undetectable viral load; 2) being unable to give informed consent; 3) Lack of Spanish language skills

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Retention in care | Six month follow up
  Retention in care will be assessed through the following measures: HIV medical care visits, ART use, self-reported adherence, acute care utilization, viral load, and health-related quality of life

SECONDARY OUTCOMES:
Intermediate outcome variables | Six month follow up
  Social support, perceived social norms, retention knowledge, retention self-efficacy, outcome expectations

CONTACTS AND LOCATIONS:
Overall Officials: William E Cunningham, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- AltaMed, Los Angeles, California, United States